CLINICAL TRIAL: NCT04833543
Title: Verticalization With Vestibular Stimulation for Patients With Severe Disorders of Consciousness: A Novel Application of a Robotic Exoskeleton
Brief Title: Verticalization Robotic Exoskeleton DoC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial Hermann Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MH-20-0834
Record Dates: First submitted 2021-03-23; First posted 2021-04-06 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Brain Injuries; Disorder of Consciousness
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tilt Table (Active Comparator)
  Interventions: Other: Tilt Table
- Robotic Mobility Device (REX) (Experimental)
  Interventions: Other: Robotic Mobility Device (REX)

INTERVENTIONS:
Other: Robotic Mobility Device (REX) — A self supporting robotic mobility device (REX) will be utilized. It is a Class I device, and it is classified as powered exercise equipment meant for anyone that requires use of a wheelchair for mobility who has difficulty with standing and walking. The participant will be supported securely within the device using a pelvic harness, and thigh and calf cuffs. The device will be operated under the supervision of a device trained physical therapist and therapy technician. The participant will be transferred into the device in a seated position. Once aligned properly and strapped in, the participant will be passively moved by the device into standing and walking positions. To provide constant vestibular input, a variety of mobility functions will be performed including standing, sitting, walking, turning, shuffling (side-stepping), and backwards stepping.
  Arms: Robotic Mobility Device (REX)
Other: Tilt Table — A tilt table is a table with a footplate that can be tilted at different angles. The participant will lie flat on the table and straps will be placed to stabilize the trunk and lower extremities. The inclination of the tilt table will be adjusted from a horizontal to a vertical position to allow the participant to attain and maintain a standing or partial-standing position. Sessions will be supervised by a physical therapist and therapy technician.
  Arms: Tilt Table

SUMMARY:
Mobilization, specifically verticalization, has been shown to play a role in enhancing consciousness. Vestibular stimulation has the potential to influence the neural substrate of consciousness, but this modality has not been thoroughly explored. The primary aim of this study is to compare the influence of verticalization with and without vestibular input on level of consciousness in patients experiencing disorders of consciousness (DoC).

ELIGIBILITY:
Inclusion Criteria:

1. unresponsive wakefulness syndrome/vegetative state (UWS/VS) or minimally conscious state (MCS) following traumatic brain injury (TBI), intracerebral bleeding, ischemic infarction, or hypoxic brain injury
2. Medical clearance by a physician
3. 18-75 years old
4. Mobilization into standing for at least 10 minutes without signs of orthostasis

Exclusion Criteria:

1. Time since injury less than 4 weeks or more than 6 months
2. Mobilization into standing lasts more than 30 minutes
3. Severe osteoporosis
4. Muscle tone that prevents joint motion (Modified Ashworth Scale (MAS) 4)
5. Unstable fractures
6. Decubiti on areas contacted by robotic mobility device (i.e. heels, tibia, greater trochanter, ischial tuberosity, sacrum)
7. Inability to fit device requirements*

   * Height 4'8"-6'4", Weight 88-222 lbs., Hip Flexion 0-90˚, Knee Flexion 0-90˚, Plantigrade

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised (CRS-R) | through study completion; an average of 8 weeks
  scores range from 0-23; higher scores mean a better outcome

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | through study completion; an average of 8 weeks
  scores range from 0-4; lower scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- TIRR Memorial Hermann, Houston, Texas, United States